CLINICAL TRIAL: NCT00956033
Title: Skin Biopsies in Chemotherapy-induced Neuropathy
Status: Completed | Type: Observational
Sponsor: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, Joost LM Jongen, J.L.M. Jongen, MD, PhD, Erasmus Medical Center
Other Study IDs: MEC2008-305
Record Dates: First submitted 2009-08-10; First posted 2009-08-11 (Estimated); Last update posted 2014-12-24 (Estimated); Status verified 2014-12

CONDITIONS: Multiple Myeloma; Peripheral Neuropathy
Keywords: Cancer; Peripheral Neuropathy; Bortezomib
MeSH Terms: conditions — Multiple Myeloma; Peripheral Nervous System Diseases; Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — skin biopsy
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with multiple myeloma

SUMMARY:
Neuropathy is a common side effect of chemotherapeutics used for the treatment of multiple myeloma, including vincristine, thalidomide and bortezomib. The neuropathy induced by these drugs is often preferentially small fiber. Small fiber neuropathies are difficult to diagnose and quantify using conventional electromyography. Determining intra-epidermal nerve fiber density (IENFD) in skin biopsies from diabetes and AIDS patients has been shown to be a more sensitive and more specific ancillary investigation to establish the diagnosis of small fiber neuropathy. In this study the investigators aim to establish the sensitivity of IENFD measurements in skin biopsies from patients with multiple myeloma treated with bortezomib.

ELIGIBILITY:
Inclusion Criteria:

* Patients with multiple myeloma receiving bortezomib

Exclusion Criteria:

* Patients not able to provide informed consent
* Patients with coagulation disturbances or immunocompromised patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with multiple myeloma receiving bortezomib in a large university hospital
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2008-11; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
intraepidermal nerve fiber density/pain intensity | one timepoint, i.e. date of skin biopsy
  correlation between intraepidermal nerve fiber density and pain intensity

CONTACTS AND LOCATIONS:
Overall Officials: Joost L Jongen, Principal Investigator — Erasmus Medical Center
Locations (1):
- Erasmus MC, Centrumlocatie en Daniel den Hoed, Rotterdam, South Holland, Netherlands

REFERENCES:
- See also: Related Info — http://www.erasmusmc.nl/neurologie